CLINICAL TRIAL: NCT03181776
Title: Hemodynamic Effect of Three Randomized Angles of Left Tilting After Spinal Anesthesia for Cesarean Delivery
Brief Title: Hemodynamic Effect of Left Tilting in Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N-36-2016
Record Dates: First submitted 2017-04-17; First posted 2017-06-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Cesarean Section Complications; Spinal Anesthetic Complications
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: The study will investigate the effect of different tilting angles on the hemodynamics of full term pregnants before and after spinal anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- left lateral tilting arm (Experimental): all patients will be put in three angles of left lateral tilt in randomized order (supine position - left lateral tilting in 15 degrees - and left lateral tilting in 30 degrees) and the hemodynamic data will be compared in the three angles.
  Interventions: Other: left lateral tilting in 15 degrees; Other: left lateral tilting in 30 degrees; Other: supine position

INTERVENTIONS:
Other: left lateral tilting in 15 degrees — The mother will be placed in left lateral tilted position (15 degrees) using a standard wedge
Other: left lateral tilting in 30 degrees — The mother will be placed in left lateral tilted position (30 degrees) using a standard wedge
Other: supine position — The mother will be placed in standard supine position

SUMMARY:
The aim of this work is to investigate the effect of different angles of lateral tilt on the maternal hemodynamics before and after subarachnoid block

DETAILED DESCRIPTION:
Aortocaval compression (ACC) by the gravid uterus is a known physiological phenomenon that is classically claimed to cause supine hypotension in full term pregnant women. ACC has been also mentioned as a possible cause of post-spinal hypotension (PSH) in parturients undergoing cesarean section (CS); however, the evidence for the value of left lateral tilting of parturient in improving hemodynamics is not clear.

The aim of this work is to investigate the effect of different angles of lateral tilt on the maternal hemodynamics before and after subarachnoid block (SAB).

Hemodynamic variables will be taken before SAB in three angles (zero angle, 15 degree angle, and 30 degree angles) of left lateral tilt.

Patients will receive normal SAB after prophylactic vasopressor adminstration (either 15 mg ephedrine or 1.5 mcg/Kg phenylephrine intravenous bolus) then hemodynamic variables will measured again after SAB in the same three angles. The sequence of the tilting angles will be randomized.

Another measure will be taken after delivery of the fetus. SAB will be done in sitting position under complete asepsis using 25 g spinal needle with crystalloid infusion of 500 mL. SAB will be achieved by intrathecal injection of 10 mg hyperbaric Bupivacaine plus 25ug fentanyl. Success of SAB will be tested within five minutes after drug injection. SAB will be considered successful if adequate block reached T4 dermatome.

Cardiac output and stroke volume will be measured using electrical cardiometry device.

ELIGIBILITY:
Inclusion Criteria:

* full term parturients scheduled for cesarean delivery

Exclusion Criteria:

* BMI > 35 Kg/m2, polyhydramnios, history of impaired cardiac contractility, valvular heart disease, cardiac arrhythmias, hypertensive pregnancy disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-11-25 (Estimated); Study Completion 2018-12-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | 30 minutes after spinal anesthesia in different angles of left lateral tilting
  Cardiac output in liters per minute measured by electrical cardiometry

SECONDARY OUTCOMES:
cardiac output | before spinal anesthesia in different angles of left lateral tilting
  Cardiac output in liters per minute measured by electrical cardiometry
mean arterial blood pressure | before spinal anesthesia in different angles of left lateral tilting
  mean arterial blood pressure measured by non-invasive monitor
mean arterial blood pressure | 30 minutes after spinal anesthesia in different angles of left lateral tilting
  mean arterial blood pressure measured by non-invasive monitor
stroke volume | before spinal anesthesia in different angles of left lateral tilting
  stroke volume in milliliters measured by electrical cardiometry
stroke volume | 30 minutes after spinal anesthesia in different angles of left lateral tilting
  stroke volume in milliliters measured by electrical cardiometry
systemic vascular resistance | before spinal anesthesia in different angles of left lateral tilting
  measured in mmHg × min / mL by electrical cardiometry
systemic vascular resistance | 30 minutes after spinal anesthesia in different angles of left lateral tilting
  measured in mmHg × min / mL by electrical cardiometry
heart rate | before spinal anesthesia in different angles of left lateral tilting
  measured in beat per minute
heart rate | 30 minutes after spinal anesthesia in different angles of left lateral tilting
  measured in beat per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No